CLINICAL TRIAL: NCT05815381
Title: Autoimmune Mechanisms in Fibromyalgia
Acronym: FMIgG
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); The Swedish Rheumatism Ass (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Eva Kosek, Professor, senior consultant, Karolinska Institutet
Other Study IDs: 2019-06161
Record Dates: First submitted 2022-11-08; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Autoimmunity; IgG antibodies; Satellite glia cells
MeSH Terms: conditions — Fibromyalgia; Autoimmune Diseases | interventions — Surveys and Questionnaires; Blood Specimen Collection; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum, skin biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia patients: Female sex, age 20-65 years and fulfilling the ACR 1990 and ACR 2016 fibromyalgia diagnostic criteria.
  Interventions: Other: Questionnaires, quantitative sensory testing, blood sampling, skin biopsies, functional magnetic resonance imaging, magnetic resonance spectroscopy
- Healthy controls: Sex and age matched healthy controls.
  Interventions: Other: Questionnaires, quantitative sensory testing, blood sampling, skin biopsies, functional magnetic resonance imaging, magnetic resonance spectroscopy

INTERVENTIONS:
Other: Questionnaires, quantitative sensory testing, blood sampling, skin biopsies, functional magnetic resonance imaging, magnetic resonance spectroscopy — se arm/group descriptions

SUMMARY:
A cohort of fibromyalgia (FM) patients (n =90) and healthy controls (HC) (n= 93) was recruited to investigate the associations between human IgG binding to satellite glia cells (SGC) from dorsal root ganglia (DRG) and pathophysiological mechanisms. The study is based on previously identified mechanisms resulting from injecting human IgG antibodies from FM patients, but not HC, in mice (Goebel et al. J Clin Invest. 2021;131(13):e144201). Subjects have been carefully phenotyped using validated questionnaires and quantitative sensory testing (QST) was applied to determine pain sensitivity. A blood sample was taken to quantify anti-SGC IgG, as well as proteins, lipids and metabolites. Skin biopsies were taken to analyze changes in skin innervation (IENFD) and immune cell activation. Magnetic resonance spectroscopy (MRS) and functional magnetic resonance imaging (fMRI) was performed (n=122) to investigate central nervous system pain related mechanisms. Insular glutamate levels, as well as the levels of other brain metabolites will be determined (MRS) and related to symptom severity and anti-SGC IgG levels. Resting state as well as pain related cerebral activation (BOLD) during standardized evoked pain stimuli will be characterized (fMRI) and related to the MRS findings and to anti-SGC IgG levels.

DETAILED DESCRIPTION:
Visit 1 (duration approx. 2,5-4 hours)

Questionnaires: A check of inclusion and exclusion criteria was made, including the palpation of tender points (ACR 1990 FM criteria). Subjects completed a set of validated questionnaires regarding pain (pain intensity ratings on visual analogue scale (VAS), pain duration, pain drawing, Short form McGill), fibromyalgia severity (fibromyalgia impact questionnaire, (FIQ)), sleep (Pittsburgh Sleep Inventory Questionnaire, (PSQI)), fatigue (Multidimensional Fatigue Inventory (MFI-20)), depression/anxiety (Hospital anxiety depression scale (HADS), Becks depression inventory (BDI), State Trait Anxiety Questionnaire (STAI)), pain coping (Coping Strategy Questionnaire (PCS)), acceptance and flexibility (chronic pain acceptance questionnaire (CPAQ-8), acceptance and action questionnaire (SAAQ)), the Tampa Scale for Kinesiophobia (TSK) and health related quality of life (EQ-5D).

Quantitative sensory testing: Perception thresholds for non-painful and painful heat/cold were examined using a Thermotest. A thermode (2x2cm) was placed at the skin and the temperature was modulated by a computer (0-50 degrees C). The subject signaled the respective perception by pressing a button, which terminated the stimulation. Subjects were instructed to press the button at the sensation of the slightest warmth/cold and when the heat/cold become painful. Sensitivity to suprathreshold heat/cold pain stimuli were determined by asking the subject to press the button when they would rate a pain intensity corresponding to 4 and 7/10. Pain sensitivity to pressure was assessed by pressure algometry at 8 different sites in the body. The subjects were instructed to press a signal button when the pressure turned into the slightest sensation of pain (pressure pain threshold) and when the pain corresponded to 4 and 7/10, respectively.

Blood test: Venous blood tests were taken (maximal volume 50 ml/individual). The levels of human IgG binding to murine satellite glia cells (SGC) will be determined as % SGC binding human IgG. In addition, we will also assess the amount of IgG binding to human DRG sections and possibly also to human SGC (postmortem donors). The blood samples will also be analysed for algogenic and inflammatory substances, lipids and metabolites and immune cell activation, including fluorescence-activated cell sorting (FACS)(in a subgroup). As an extension of the study, IgG antibodies will be purified to evaluate the effect on cell cultures and in the rodent FM model.

Skin biopsies: Two punch skin biopsies (4 mm diameter) were performed at the thigh. The skin was sterilized, and anesthetized using a local anesthetic (10mg/ml Xylocain with adrenalin). If needed the was treated with spongostan/BloodStop and a special plaster (Steri-Strip) was always applied for 7-10 days. The skin will be analyzed regarding morphological changes of intradermal small fibres and IENFD and thick myelinated fibers will be determined. In addition, immune cell activation will be assessed using various methods.

Visit 2 (duration approx. 1,5 hours)

Imaging: The subjects were asked to make a new pain rating (VAS). They were familiarized with the evoked pain stimulus used in the scanner. Following the safety routines to exclude contraindications for MR scanning the subjects were placed in the scanner. The assessment started with structural scans (T1, T2), followed by resting state and MR spectroscopy (anterior and posterior insula) and finally an evoked pain protocol using a series of painful pressure stimuli generated by an automatic pressure applicator at the leg of the subjects, corresponding to 150 and 300kPa, respectively, (blood oxygenation level dependent, BOLD).

Aims not specified elsewhere:

1. To run assays aiming at identifying the antigen/antigens and if successful to quantify the specific antibodies and relate them to FM severity.
2. To assess if IgG antibodies form individuals with severe FM activate satellite cell cultures to release pro-inflammatory and algesic substances more efficiently than IgG antibodies from individuals with less severe FM.
3. To investigate if there are abnormalities in the number, characteristics, or activation of immune cells in the blood or skin of FM patients compared to HC.
4. To assess effects of FM IgG on animal models.

ELIGIBILITY:
Inclusion Criteria:

* Female sex,
* age 20-65 years

For the FM arm:

* fulfilling the ACR 1990 fibromyalgia diagnostic criteria
* fulfilling the ACR 2016 fibromyalgia diagnostic criteria

Exclusion Criteria:

* autoimmune or inflammatory diseases (other than FM in the FMS cohort)
* other somatic diseases that could influence the study outcome (e.g. peripheral neuropathy etc)
* pain problems (other than FM in the FMS cohort)
* severe depression/anxiety that requires specific treatments
* medication with anticonvulsants, antidepressants or corticosteroids
* inability to refrain from NSAIDs, analgesics, sedatives or sleep medication 48 hours before examinations
* inability to communicate in Swedish or other factors that the investigator judges would interfere with the participation in the study
* smoking > 5 cigarettes/day
* pregnancy
* drug or alcohol abuse
* contraindications to skin biopsy (allergy to local anesthetics, hemophilia, medication with anticoagulants)
* contraindications to fMRI (metal implants, pacemaker)

Ages: 20 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited by advertising in daily press and social media. All subjects will be pre-screened by a telephone interview from our research nurse regarding inclusion and exclusion criteria before invited to the first visit. All subjects will have to sign informed consent before being included.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Group differences in anti-SGC IgG levels | 2 years
  Difference in percent satellite glia cells bound by IgG (anti-SGC IgG levels, 0-100%, 100% worst) between fibromyalgia patients and healthy controls
Resting state cerebral activity and anti-SGC IgG levels in FM | 2 years
  Difference in resting state functional magnetic resonance imaging (exploratory approach) between fibromyalgia (FM) patients with high (50% or more) and low (less than 50%) percent satellite glia cells bound by IgG (anti-SGC IgG levels)
Cerebral activation during pressure pain (150kPa) and anti-SGC IgG levels in FM | 2 years
  Difference in blood oxygenation level dependent functional magnetic resonance imaging during evoked pain (150 kPa) between fibromyalgia (FM) patients with high (50% or more) and low (less than 50%) percent satellite glia cells bound by IgG (anti-SGC IgG levels)
Cerebral activation during pressure pain (300kPa) and anti-SGC IgG levels in FM | 2 years
  Difference in blood oxygenation level dependent functional magnetic resonance imaging during evoked pain (300 kPa) between fibromyalgia (FM) patients with high (50% or more) and low (less than 50%) percent satellite glia cells bound by IgG (anti-SGC IgG levels)
Glutamate concentrations in anterior insula and anti-SGC IgG levels in FM | 2 years
  Difference in glutamate levels, magnetic resonance spectroscopy of anterior insula, between fibromyalgia (FM) patients with high (50% or more) and low (less than 50%) percent satellite glia cells bound by IgG (anti-SGC IgG levels)
Glutamate concentrations in posterior insula and anti-SGC IgG levels in FM | 2 years
  Difference in glutamate levels, magnetic resonance spectroscopy of posterior insula between fibromyalgia (FM) patients with high (50% or more) and low (less than 50%) percent satellite glia cells bound by IgG (anti-SGC IgG levels)
Cerebral metabolites in anterior insula and anti-SGC IgG levels in FM | 2 years
  Differences in magnetic resonance spectroscopy of anterior insula between fibromyalgia (FM) patients with high (50% or more) and low (less than 50%) percent satellite glia cells bound by IgG (anti-SGC IgG levels)(exploratory)
Cerebral metabolites in posterior insula and anti-SGC IgG levels in FM | 2 years
  Differences in magnetic resonance spectroscopy of posterior insula between fibromyalgia (FM) patients with high (50% or more) and low (less than 50%) percent satellite glia cells bound by IgG (anti-SGC IgG levels)(exploratory)

SECONDARY OUTCOMES:
Group differences in resting state functional magnetic resonance imaging | 2 years
  Difference in resting state functional magnetic resonance imaging (exploratory approach) between fibromyalgia patients and healthy controls
Group differences in fMRI BOLD during evoked pressure pain (150 kPa) | 2 years
  Difference in blood oxygenation level dependent (BOLD) functional magnetic resonance imaging during evoked pain (150 kPa) between fibromyalgia patients and healthy controls
Group differences in fMRI BOLD during evoked pressure pain (300 kPa) | 2 years
  Difference in blood oxygenation level dependent functional magnetic resonance imaging during evoked pain (300 kPa) between fibromyalgia patients and healthy controls
Group differences in glutamate levels in anterior insula | 2 years
  Difference in glutamate levels, magnetic resonance spectroscopy of anterior insula, between fibromyalgia patients and healthy controls
Group differences in glutamate levels in posterior insula | 2 years
  Difference in glutamate levels, magnetic resonance spectroscopy of posterior insula, between fibromyalgia patients and healthy controls
Group differences in cerebral metabolites in anterior insula | 2 years
  Differences in magnetic resonance spectroscopy of anterior insula between fibromyalgia patients and healthy controls (exploratory)
Group differences in cerebral metabolites in posterior insula | 2 years
  Differences in magnetic resonance spectroscopy of posterior insula between fibromyalgia patients and healthy controls (exploratory)
Correlations between glutamate in anterior insula and anti-SGC IgG levels in FM | 2 years
  Spearman correlations (0-1, 1 best correlation) between glutamate levels in anterior insula, magnetic resonance spectroscopy, and percent satellite glia cells bound by IgG (anti-SGC IgG levels, 0-100%, 100% worst) in fibromyalgia (FM) patients
Correlations between glutamate in posterior insula and and anti-SGC IgG levels in FM | 2 years
  Spearman correlations (0-1, 1 best correlation) between glutamate levels in posterior insula, magnetic resonance spectroscopy, and percent satellite glia cells bound by IgG (anti-SGC IgG levels, 0-100%, 100% worst) in fibromyalgia (FM) patients
Correlations between % SGC IgG and pain intensity in FM | 2 years
  Spearman correlations (0-1, 1 best correlation) in fibromyalgia (FM) patients between percent satellite glia cells bound by IgG (% SGC IgG, range 0-100%, 100% worst) and pain intensity assessed by visual analogue scale (VAS, range 0-100, 100 worst)
Correlations between % SGC IgG and fibromyalgia severity | 2 years
  Spearman correlations (0-1, 1 best correlation) in fibromyalgia (FM) patients between percent satellite glia cells bound by IgG (% SGC IgG, range 0-100%, 100% worst) and fibromyalgia impact questionnaire (FIQ, range 0-100%, 100% most severe fibromyalgia)
Correlations between % SGC IgG and sensitivity to pressure pain in FM | 2 years
  Spearman correlations (0-1, 1 best correlation) in fibromyalgia (FM) patients between percent satellite glia cells bound by IgG (% SGC IgG, range 0-100%, 100% worst) and pressure pain sensitivity (pressure algometry, 0-1500kPa, 1500 kPa least pain sensitive)

OTHER OUTCOMES:
Correlations between % SGC IgG and IENFD | 2 years
  Spearman correlations (0-1, 1 best correlation) between percent satellite glia cells bound by IgG (% SGC IgG) and intraepidermal nerve fiber density (IENFD)(subgroup of fibromyalgia patients n= 30 and healthy controls n =30)
Correlations between IENFD and glutamate in anterior insula | 2 years
  Spearman correlations (0-1, 1 best correlation) between intraepidermal nerve fiber density (IENFD) and glutamate concentrations in anterior insula (subgroup of fibromyalgia patients n= 30 and healthy controls n = 30)
Correlations between IENFD and glutamate in posterior insula | 2 years
  Spearman correlations (0-1, 1 best correlation) between intraepidermal nerve fiber density (IENFD) and glutamate concentrations in posterior insula (subgroup of fibromyalgia patients n= 30 and healthy controls n = 30)
Correlations between % SGC IgG and sensitivity to cold pain in FM | 2 years
  Spearman correlations (0-1, 1 best correlation) in fibromyalgia (FM) patients between percent satellite glia cells bound by IgG (% SGC IgG, range 0-100%, 100% worst) and cold pain sensitivity (MSA Thermal Stimulator, 32-0 degrees Celsius, 0 degrees least pain sensitive)
Correlations between % SGC IgG and sensitivity to heat pain in FM | 2 years
  Spearman correlations (0-1, 1 best correlation) in fibromyalgia (FM) patients between percent satellite glia cells bound by IgG (% SGC IgG, range 0-100%, 100% worst) and heat pain sensitivity (MSA Thermal Stimulator, 32-50 degrees Celsius, 50 degrees least pain sensitive)
Group differences in pressure pain sensitivity | 2 years
  Differences in pressure pain sensitivity (pressure algometry, 0-1500kPa, 1500kPa least pain sensitive) between fibromyalgia patients and healthy controls
Group differences in cold pain sensitivity | 2 years
  Differences in cold pain sensitivity (MSA Thermal Stimulator, 32-0 degrees Celsius, 0 degrees least pain sensitive) between fibromyalgia patients and healthy controls
Group differences in heat pain sensitivity | 2 years
  Differences in heat pain sensitivity (MSA Thermal Stimulator, 32-50 degrees Celsius, 50 degrees least pain sensitive) between fibromyalgia patients and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kosek, Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Insitutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No